CLINICAL TRIAL: NCT02839239
Title: Role of Lactobacillus Rhamnosus (FloraActive™) 19070 and Lactobacillus Reuteri (FloraActive™) DSM 12246 in Infant Colic: a Controlled Dietary Study
Brief Title: Lactocare Baby Drops in Infants Colic
Acronym: LACONIC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Biocare Copenhagen A/S (Industry)
Collaborators: Lviv National Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IC-SVG-P0001
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: Infant Colic
MeSH Terms: conditions — Colic | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Drops with lactobacilli and vitamin D3 (Experimental): Exclusive breast feeding plus L. rhamnosus 19070-2 and L. reuteri DSM 12246 in a dose of 125 x 106 CFU (both strains) with 1,667 mg fructooligosaccharides and 2,5 mcg (100 IU) vitamin D3 (in sunflower oil) per 6 drops. One dose (6 drops) in the first morning (from 6 AM) breastfeeding, and one dose (6 drops) in one of the evening (6 PM-12 PM) breast feedings for 28 days.
  Interventions: Dietary Supplement: Drops with lactobacilli and vitamin D3
- Drops with vitamin D3 (Placebo Comparator): Exclusive breast feeding plus 2.5 mcg (100 IU) vitamin D3 (in sunflower oil) per 6 drops. One dose (6 drops) in the first morning (from 6 AM) breastfeeding, and one dose (6 drops) in one of the evening (6 PM-12 PM) breast feedings for 28 days.
  Interventions: Dietary Supplement: Drops with vitamin D3

INTERVENTIONS:
Dietary Supplement: Drops with lactobacilli and vitamin D3 — Oil suspension with lactobacilli and vitamin D3
  Arms: Drops with lactobacilli and vitamin D3
Dietary Supplement: Drops with vitamin D3 — Oil suspension with vitamin D3
  Arms: Drops with vitamin D3

SUMMARY:
The objective of this study is to determine an efficacy of the combination of L. rhamnosus 19070-2 (FloraActiveTM) and L. reuteri DSM 122460 (FloraActiveTM) in decreasing cry/fuss in infants aged 4 through 12 weeks with IC. The active group of infants will receive lactobacilli with vitamin D3 while the control group will receive vitamin D3 2 times daily as oil suspension for 28 days. Duration of infant fuss/cry will be measured at baseline and at the end of intervention to define a difference between the groups

DETAILED DESCRIPTION:
There is accumulating interest in role of lactobacilli in decreasing cry and fuss in infant colic, the condition that affects around 1 of 4-5 infants. The interest for dietary supplementation has been evoked by a line of earlier studies, indicating that infants with colic had an increased number of gas-forming E.coli in the intestines and potential interference between lactobacilli and E.coli. Systematic review of evidence, based on the 6 randomized controlled dietary studies, conducted in Italy, Poland, Australia, Canada, and Finland, has concluded of the decrease of the mean time cry of infant by -55 minutes a day after the 3 weeks dietary course with lactobacilli . In the mentioned studies most commonly used lactobacilli were L. reuteri, however, the effect of combination of L. reuteri with other lactobacilli remains unknown.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent form signed by both parents.
2. Gender: males and females;
3. Age: 4 -12 weeks;
4. Infant colic, defined as cry/fussing lasting > 3 h, occurring > 3 d for 7 days;
5. Gestational age 37-42 weeks;
6. Birth weight 2,500-4,200 g;
7. Stated availability throughout the study period;
8. Sated availability of mobile phone or phone with answering machine.

Exclusion Criteria:

1. Any formula feeding in any amount;
2. Failure to thrive (weight gain less than 100 grams per week as averaged from the birth weight to the weight at entry);
3. Current maternal smoking;
4. Known moderate or severe disease of any systems (neural, skeletal, muscular, cutaneous, gastrointestinal, respiratory, genital, urinary, immune);
5. Present intake of antibiotics by infant or mother;
6. Present intake of prebiotics or probiotics by infant or mother;
7. Difficulty of parents to comprehend study requirements as judged by the physician;
8. Suspected parental alcohol or drug addiction as judged by the physician.

Ages: 4 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 168 (Actual)
Dates: Start 2016-12-09; Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Change in mean cry/fuss time (min/day) from day 0 through day 28 | 28 days
  Change in mean cry/fuss time

SECONDARY OUTCOMES:
Change in mean cry time (min/day) from day 0 through day 28 | 28 days
  Change in mean cry time
Change in mean fuss time (min/day) from day 0 through day 28 | 28 days
  Change in mean fuss time
Treatment success (percent) at 7, 14, 21, 28 days, defined as more than 25% and 50% reduction in cry time from baseline | 7, 14, 21, 28 days
  Outcome Measure Description
Recovery success (percent) at 7, 14, 21, 28 days, defined as reduction in duration of cry time less than 3 hours per day (unmet Wessel criteria); | 7, 14, 21, 28 days
  Recovery success
Cry and fuss time (min/day) on days 0, 7, 14, 21, 28 | 7, 14, 21, 28 days
  Cry and fuss time

OTHER OUTCOMES:
Infant sleep duration (min/day) on days 0, 7, 14, 21, 28 | 7, 14, 21, 28 days
  Infant sleep duration
Change in maternal depression score from day 0 through day 28 | 28 days
  Change in maternal depression score

CONTACTS AND LOCATIONS:
Overall Officials: Soren Thomsen, Study Director — Biocare Copenhagen A/S

IPD SHARING:
Plan to Share IPD: Undecided